CLINICAL TRIAL: NCT01907529
Title: A Trail of Neoadjuvant Endostar in Combination With Docetaxel, Epirubicin and Cyclophosphamide in Patients With Stage III Breast Cancer (TENDENCY)
Brief Title: A Trail of Neoadjuvant Endostar in Combination With Chemotherapy in Breast Cancer
Acronym: TENDENCY
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Hebei Medical University Fourth Hospital (Other)
Responsible Party: Principal Investigator, Yunjiang Liu, M.D, Chief Physician of Breast Cancer Dept, Vice-President of Hebei Medical University Fourth Hospital, Hebei Medical University Fourth Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HBMUFH-101
Record Dates: First submitted 2013-07-22; First posted 2013-07-25 (Estimated); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Stage III Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Epirubicin; Cyclophosphamide; endostar protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemo plus Endostar (Experimental): Docetaxel, epirubicin and cyclophosphamide plus endostar
  Interventions: Drug: docetaxel, epirubicin and cyclophosphamide plus endostar
- Chemo only (Active Comparator): docetaxel, epirubicin and cyclophosphamide
  Interventions: Drug: docetaxel, epirubicin and cyclophosphamide

INTERVENTIONS:
Drug: docetaxel, epirubicin and cyclophosphamide — docetaxel 75mg/m2, IV (in the vein) on day 1 of each 21 day cycle; epirubicin 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle, cyclophosphamide 500mg/m2, IV (in the vein) on day 1 of each 21 day cycle; totally 4 cycles
  Arms: Chemo only
Drug: docetaxel, epirubicin and cyclophosphamide plus endostar — docetaxel 75mg/m2, IV (in the vein) on day 1 of each 21 day cycle; epirubicin 75 mg/m2, IV (in the vein) on day 1 of each 21 day cycle, cyclophosphamide 500mg/m2, IV (in the vein) on day 1 of each 21 day cycle; endostar 7.5mg/m2, IV (in the vein) from day 1 to day 14, totally 4 cycles
  Arms: Chemo plus Endostar

SUMMARY:
The trial was designed to study the efficacy and safety of neoadjuvant docetaxel, epirubicin in combination with cyclophosphamide(DEC) plus human recombinant endostatin (endostar) for breast cancer patients. The hypothesis of this protocol is that the combined an active angiogenesis agent to chemotherapy could enhance the pathological responce rate and further benefit breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed invasive breast cancer (core needle biopsy for breast cancer diagnosis and fine needle aspiration for lymph node metastasis diagnosis)
* Age 18-70
* No evidence of distant metastasis
* No previous therapy
* Normal hematologic function
* No abnormality of renal or liver function
* Written informed consent

Exclusion Criteria:

* With allergic constitution or possible allergic reflection to drugs to be used in this study
* Any concurrent uncontrolled medical or psychiatric disorder
* History of severe heart diseases, including congestive heart failure, unstable angina, uncontrolled arrhythmia, myocardial infarction, uncontrolled high blood pressure, or heart valve disease
* Being pregnant or nursing

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2020-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Clinical/pathological response | 48 months
  The clincial response will be evaluated according to RECIST criteria.

SECONDARY OUTCOMES:
PFS | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: YUNJIANG LIU, M.D.& PhD., Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- Fourth Hospital of Hebei Medical University, Tumor Hospital of Hebei Province, China, Shijiazhuang, Hebei, China